CLINICAL TRIAL: NCT00373828
Title: Non-cardiac Chest Pain Evaluation and Treatment Study (CARPA) - Part 1: Diagnosis
Status: Completed | Type: Observational
Sponsor: Clinical Locomotion Science (Other)
Collaborators: Nordic Institute of Chiropractic and Clinical Biomechanics (Other); Odense University Hospital (Other); University of Southern Denmark (Other); The County of Funen, Denmark (Other Government); Foundation for Chiropractic Research and Post Graduate Education (Other)
Responsible Party: Principal Investigator, Mette Jensen Stochkendahl, DC, PhD, Clinical Locomotion Science
Other Study IDs: Project 73 (NUA)
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Non-Cardiac Chest Pain; Undiagnosed Chest Pain; Musculoskeletal Chest Pain; Ischemic Heart Disease
Keywords: Chest Pain; Chest Wall; Angina Pectoris; Atypical Chest Pain; Physical Examination; Myocardial Perfusion Imaging; Observational Study; Non-Cardiac Chest Pain; Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia; Chest Pain; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The overall aim of the project is to evaluate diagnosis and treatment of chest pain originating from the musculoskeletal system. Specifically, we wish to investigate prevalence and character of such chest pain in a population of patients with acute chest pain, admitted to a university hospital based acute chest pain clinic, and undergoing evaluation of acute coronary syndrome (Part 1). Then, to test a manually-based treatment protocol to patients with diagnosed musculoskeletal chest pain in a randomized clinical trial (Part 2).

The specific purpose of this study (Part 1) is to determine the exact number of patients with acute chest pain origination from the musculoskeletal system, and to describe their cardiac status with respect to ischemic heart disease. Further, we wish to evaluate the decision making process of the chiropractor.

DETAILED DESCRIPTION:
Acute chest pain is a common reason for hospital admission. The focus of diagnosis is of course pain of cardiac origin including myocardial infarction and/or other ischemic heart disease; however, in up to 50% of cases the aetiology may be non-cardiac. Differential diagnoses include primarily pulmonary, gastrointestinal, psychosocial, or musculoskeletal problems, and musculoskeletal problems may account for around 20% of the total number of admissions in acute chest pain clinics. Thus the musculoskeletal system is a recognized possible source of pain in patients with chest pain even though a confident diagnosis of musculoskeletal chest pain can be difficult to establish since no gold standard exists to verify this diagnosis.

Chest pain patients with normal coronary anatomy have an excellent prognosis for survival and a future risk of cardiac morbidity similar to that reported in the background population. However, about three quarters of patients with non-cardiac chest pain continue to suffer from residual chest pain with large socio-economic consequences. Therefore, a search for an alternative cause with related possibilities for treatment is warranted. Given these perspectives, the general objective of the present work is to study the diagnosis of chest pain originating from the musculoskeletal system of the cervical and thoracic spine, and thorax in patients with chest pain of various origins, and to evaluate ischemic heart disease status among patients with presumed musculoskeletal pain.

Evaluation:

Patients with musculoskeletal chest pain will be identified using a standardized examination protocol comprised of a semi-structured interview, a general health examination, and a specific manual examination of the muscles and joints of the neck, thoracic spine and thorax. All patients will have a Myocardial Perfusion Imaging (MPI) performed and results from the MPI will be compared with the musculoskeletal status. Specific important parameters of the standardized examination protocol will be identified and the decision making process of the chiropractor will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Acute episode of chest pain of less than 7 days duration as primary reason for admission to a chest pain clinic.
* Admitted to a chest pain clinic, suspected of acute coronary infarction, but with a negative diagnosis confirmed by normal coronary enzymes and normal ECG.
* Pain arising from the thorax and/or neck.
* Able to read and understand Danish.

Exclusion Criteria:

* Acute coronary syndrome.
* Percutaneous Coronary Intervention.
* Coronary Artery Bypass Grafting.
* Other disease, diagnosed during this admission, which is likely to have caused the acute episode of chest pain.
* No written consent.
* Inflammatory joint disease.
* Diabetes mellitus, type I.
* Fibromyalgia.
* Sharp trauma to the chest.
* Malignant disease.
* Apoplexy.
* Gross osseous anomalies, such as pronounced scoliosis.
* Known or suspected osteoporosis.
* Pregnancy.
* Dementia/unable to cooperate.
* Not residing in the County of Funen.
* Does not want to participate.
* Other - reason for exclusion will be noted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three hundred consecutive patients with an episode of suspected non-cardiac acute chest pain will be recruited from among patients discharged from an acute chest pain clinic situated at a large specialized cardiology department.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2006-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal chest pain | baseline
  Presence of MSCP yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Poul Flemming Hoilund-Carlsen, Professor, Study Chair — The Dept. of Nuclear Medicine, Odense University Hospital; Torben Haghfelt, Professor, Study Chair — The Dept. of Cardiology, Odense University Hospital
Locations (1):
- The Dept. of Cardiology and Dept. of Nuclear Medicine, Odense University Hospital, Sdr. Boulevard 29, Odense C, Denmark

REFERENCES:
- [Background] Stochkendahl MJ, Christensen HW, Vach W, Hoilund-Carlsen PF, Haghfelt T, Hartvigsen J. Diagnosis and treatment of musculoskeletal chest pain: design of a multi-purpose trial. BMC Musculoskelet Disord. 2008 Mar 31;9:40. doi: 10.1186/1471-2474-9-40. PMID 18377636
- [Result] Stochkendahl MJ, Vach W, Hartvigsen J, Hoilund-Carlsen PF, Haghfelt T, Christensen HW. Reconstruction of the decision-making process in assessing musculoskeletal chest pain: an exploratory study using recursive partitioning. J Manipulative Physiol Ther. 2012 Mar-Apr;35(3):184-95. doi: 10.1016/j.jmpt.2012.01.009. Epub 2012 Feb 27. PMID 22377444
- See also: Related Info — http://www.nikkb.dk